CLINICAL TRIAL: NCT00909909
Title: Safety and Feasibility of Accelerated, Hypofractionated Radiotherapy in Women With Breast Cancer: A Phase II Trial
Brief Title: Radiation Therapy in Treating Women With Early Stage Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, Bruce G Haffty, Professor and Chairman, Department of Radiation Oncology, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro20170001671; CDR0000643276 (Other: NIH); P30CA072720 (NIH); 0220090059 (Other: IRB); 040807 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ; invasive ductal breast carcinoma; invasive lobular breast carcinoma; medullary ductal breast carcinoma with lymphocytic infiltrate; mucinous ductal breast carcinoma; papillary ductal breast carcinoma; tubular ductal breast carcinoma; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Carcinoma, Ductal, Breast; Carcinoma, Lobular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): 3DCRT/IMRT lumpectomy bed boost followed by accelerated whole breast irradiation (AWBI)
  Interventions: Radiation: External beam boost; Radiation: whole breast irradiation
- B (Active Comparator): Accelerated whole breast irradiation (AWBI) followed by 3DCRT/IMRT lumpectomy bed boost
  Interventions: Radiation: External beam boost; Radiation: whole breast irradiation

INTERVENTIONS:
Radiation: External beam boost — 3-dimensional conformal radiation therapy and intensity modulated radiation therapy
Radiation: whole breast irradiation — accelerated, hypofractionated whole breast irradiation

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy in different ways may kill more tumor cells. Giving it after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying the side effects of radiation therapy and to see how well it works in treating women with early stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the freedom from local and regional failure in women with early stage breast cancer treated with accelerated, hypofractionated radiotherapy.
* To determine the acute and late toxicity of accelerated, hypofractionated radiotherapy using previously published toxicity scales.

Secondary

* To measure cosmesis using the Harvard cosmesis scale in patients who have undergone lumpectomy.
* To identify co-variates responsible for poor cosmetic outcome in these patients.

OUTLINE: Patients who have undergone lumpectomy undergo either intracavitary balloon brachytherapy boost and hypofractionated, accelerated whole breast irradiation (AWBI) OR 3D-conformal radiotherapy (3D-CRT)/intensity-modulated radiotherapy (IMRT) boost and AWBI. Patients who have undergone mastectomy undergo hypofractionated, accelerated chest wall irradiation.

* Intracavitary balloon brachytherapy boost and AWBI (post-lumpectomy): Patients undergo intracavitary balloon brachytherapy boost twice daily for 2 days (total of 4 fractions). Beginning 5-21 days after completion of brachytherapy, patients undergo AWBI once daily 5 days a week for approximately 2 weeks (total of 11 fractions).
* 3D-CRT/IMRT boost and AWBI (post-lumpectomy): Patients undergo 3D-CRT/IMRT boost twice daily for 2 days (total of 4 fractions). Patients also undergo AWBI as above before or after boost radiotherapy.
* Accelerated chest wall irradiation (post-mastectomy): Patients undergo accelerated chest wall irradiation once daily 5 days a week for approximately 2 weeks (total of 11 fractions).

Patients who have undergone lumpectomy undergo frontal digital photography of the breasts at baseline, immediately before the initiation of radiotherapy, and then annually for 3 years after completion of radiotherapy. These patients also complete the Breast Cancer Treatment Outcome Scale at baseline and at 3 years after completion of radiotherapy. Physicians complete the Harvard Cosmesis scale at baseline and at 1 and 3 years after completion of radiotherapy.

After completion of study treatment, patients are followed up at weeks 1, 4, and 8 and then every 4 months for 2 years, every 6 months for 3 years, and annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer, including 1 of the following subtypes:

  * Ductal carcinoma in situ
  * Invasive ductal carcinoma
  * Invasive lobular carcinoma
  * Medullary carcinoma
  * Papillary carcinoma
  * Colloidal (mucinous) carcinoma
  * Tubular carcinoma
* Pathological stage 0-IIIA disease (pTis; pT1-2, N0-N2a, M0)

  * Tumor size ≤ 5 cm
* Breast considered technically satisfactory for radiotherapy
* Has undergone lumpectomy or mastectomy and either sentinel node biopsy or axillary dissection (if invasive carcinoma is present)

  * Negative inked histological margins (i.e., no invasive cells at surgical margin) or confirmed negative re-excision specimen
* Unifocal or multifocal (confined to 1 quadrant; tumors < 4 cm apart) disease with 1 or 2 foci that can be encompassed by 1 lumpectomy
* No proven multicentric carcinoma (tumors in different quadrants of the breast or tumor separated by ≥ 4 cm) with other clinically or radiographically suspicious areas in the ipsilateral breast unless confirmed to be negative for malignancy by biopsy
* No evidence of suspicious microcalcifications in the breast before the start of radiotherapy

  * If malignancy-associated microcalcifications were initially present, the post-excision mammography must be negative
* No more than 9 positive axillary lymph nodes
* No palpable or radiographically suspicious contralateral axillary, supraclavicular, infraclavicular, or internal mammary nodes unless there is histologic confirmation that these nodes are negative for tumor
* No previously treated contralateral breast cancer or synchronous ipsilateral breast cancer
* No lobular carcinoma in situ alone (i.e., no invasive component) or non-epithelial breast malignancies (e.g., sarcoma or lymphoma)
* No Paget disease of the nipple
* No skin involvement, regardless of tumor size
* No distant metastases
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Pre- or post-menopausal
* ECOG performance status 0-1
* No co-existing medical condition that would limit life expectancy to < 2 years
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except for nonmelanoma skin cancer (the disease-free interval from any prior malignancy must be continuous)
* No collagen vascular disease, specifically systemic lupus erythematosus, scleroderma, or dermatomyositis
* No psychiatric or addictive disorder that would preclude obtaining informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy for the current breast cancer
* No tylectomies so extensive that the cosmetic result is low or poor prior to radiotherapy
* Chemotherapy allowed provided the following criteria are met:

  * Chemotherapy is not administered prior to, during, and for ≥ 21 days after completion of radiotherapy (for patients receiving brachytherapy boost)
  * Chemotherapy is not administered for ≥ 21 days before, during, and for ≥ 21 days after completion of radiotherapy (for patients receiving external beam radiotherapy boost or chest wall irradiation)
* Concurrent tamoxifen, anastrozole, or other hormonal therapy allowed

  * May be initiated before, during, or after radiotherapy
* No other concurrent chemotherapy, immunotherapy, or experimental medications

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-05-13 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Loco-regional control as assessed by physical examination, mammography, and other relevant imaging | 5 years

SECONDARY OUTCOMES:
Toxicity (including seroma formation, brachial plexopathy, fat necrosis, pain, pigmentation, and telangiectasia) as assessed by NCI CTCAE v3.0 | 5 years
Cosmesis as assessed by the Breast Cancer Treatment Outcome Scale | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Haffty, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (4):
- United States (4):
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, Hamilton, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, Somerset, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chakraborty MA, Sherwani ZK, Narra LR, Abou Yehia Z, Ohri N, Cui T, Eladoumikdachi F, Kowzun MJ, Kumar S, Potdevin L, Toppmeyer DL, Haffty BG. Preoperative Radiation Boost Results in Low Rates of Re-excision and Reduced Locoregional Treatment Time in Breast Cancer Patients. Ann Surg Oncol. 2025 Dec;32(13):9836-9842. doi: 10.1245/s10434-025-18089-9. Epub 2025 Aug 20. PMID 40836156
- [Derived] Ahlawat S, Haffty BG, Goyal S, Kearney T, Kirstein L, Chen C, Moore DF, Khan AJ. Short-Course Hypofractionated Radiation Therapy With Boost in Women With Stages 0 to IIIa Breast Cancer: A Phase 2 Trial. Int J Radiat Oncol Biol Phys. 2016 Jan 1;94(1):118-125. doi: 10.1016/j.ijrobp.2015.09.011. Epub 2015 Sep 16. PMID 26700706